CLINICAL TRIAL: NCT01215669
Title: Immunogenicity and Safety of Sanofi Pasteur's Intradermal Influenza Vaccine (IDflu™) in Adults and Elderly in Korea
Brief Title: Study of Sanofi Pasteur's Intradermal Influenza Vaccine (IDflu™) in Adults and Elderly in Korea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GID33; U111111156473 (Other: WHO)
Record Dates: First submitted 2010-10-05; First posted 2010-10-06 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Influenza
Keywords: Influenza; Influenza Virus Vaccines; Intradermal Injections
MeSH Terms: conditions — Influenza, Human | interventions — vaxigrip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: Adult Intradermal (ID) Vaccine (Experimental): Participants aged 18 to 59 years will be vaccinated with IDflu™ influenza vaccine
  Interventions: Biological: IDflu™: Split virion inactivated influenza vaccine
- Group 2: Adult Intramuscular (IM) Vaccine (Active Comparator): Participants aged 18 to 59 years will be vaccinated with Vaxigrip® Influenza vaccine
  Interventions: Biological: Vaxigrip®: Split virion inactivated influenza vaccine
- Group 3: Elderly Intradermal (ID) Vaccine (Experimental): Participants aged 60 years or older will be vaccinated with IDflu™ Influenza vaccine
  Interventions: Biological: IDflu™: Split virion inactivated influenza vaccine
- Group 4: Elderly Intramuscular (IM) Vaccine (Active Comparator): Participants aged 60 years or older will be vaccinated with Vaxigrip® Influenza vaccine
  Interventions: Biological: Vaxigrip®: Split virion inactivated influenza vaccine

INTERVENTIONS:
Biological: IDflu™: Split virion inactivated influenza vaccine — Single dose 0.1 mL, intradermal
  Other Names: IDflu™
  Arms: Group 1: Adult Intradermal (ID) Vaccine
Biological: Vaxigrip®: Split virion inactivated influenza vaccine — Single dose 0.5 mL, intramuscular
  Other Names: Vaxigrip®
  Arms: Group 2: Adult Intramuscular (IM) Vaccine
Biological: IDflu™: Split virion inactivated influenza vaccine — Single dose 0.1 mL, intradermal
  Other Names: IDflu™
  Arms: Group 3: Elderly Intradermal (ID) Vaccine
Biological: Vaxigrip®: Split virion inactivated influenza vaccine — Single dose 0.5 mL, intramuscular
  Other Names: Vaxigrip®
  Arms: Group 4: Elderly Intramuscular (IM) Vaccine

SUMMARY:
This study is designed to assess the immunogenicity and safety of the 2010-2011 NH season formulation of intradermal (ID) influenza vaccine as part of a post registration commitment.

Objectives:

* For all groups, to evaluate compliance, in terms of immunogenicity, of the corresponding strength of the intradermal (ID) or intramuscular (IM) influenza vaccine Northern Hemisphere (NH) 2010 2011 formulation with the requirements of the Committee for Human Medicinal Products (CHMP) Note for Guidance (NfG) CPMP/BWP/214/96
* For all groups, to describe the safety

DETAILED DESCRIPTION:
All participants will receive a single dose of study vaccine on Day 0. Immunogenicity data will be collected before vaccination and on Day 21 post vaccination. Safety will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman of childbearing potential, use of an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination.

Exclusion Criteria:

* Known systemic hypersensitivity to eggs, chicken proteins, neomycin, formaldehyde and octoxynol-9, or to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Known pregnancy, or a positive urine pregnancy test
* Currently breastfeeding a child
* History of seasonal influenza vaccination within the previous 6 months (other than pandemic H1N1 influenza vaccine)
* Receipt of an influenza vaccine (either seasonal or pandemic vaccine) in a clinical trial within the previous 12 months
* Known or suspected congenital or acquired immunodeficiency, resulting for example from: end-stage renal disease requiring dialysis; active neoplastic disease or active hematologic malignancy; receipt of immunosuppressive therapy or other immune-modifying drugs such as, but not limited to anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* History of seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* History of thrombocytopenia, contraindicating intramuscular (IM) vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination, under the investigator's judgment
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination
* Planned receipt of any vaccine in the 3 weeks following the trial vaccination
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Identified as employees of the Investigator or study department, with direct involvement in the proposed study or other studies under the direction of that Investigator or study department as well as family members (i.e., immediate, husband, wife and their children, adopted or natural) of the employees or the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Information concerning the immunogenicity of intradermal influenza vaccine in terms of seroprotection status (titers ≥40) using the Hemagglutination Inhibition (HAI) technique. | 21 days post-vaccination
Information regarding the safety (in terms of solicited injection site and systemic reactions) post-vaccination | Day 0 to up to 21 days post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (1):
- Seoul, South Korea

REFERENCES:
- [Result] Hoon Han S, Hee Woo J, Weber F, Joo Kim W, Ran Peck K, Il Kim S, Hwa Choi Y, Myung Kim J. Immunogenicity and safety of Intanza((R))/IDflu((R)) intradermal influenza vaccine in South Korean adults: a multicenter, randomized trial. Hum Vaccin Immunother. 2013 Sep;9(9):1971-7. doi: 10.4161/hv.25295. Epub 2013 Jun 18. PMID 23778938